CLINICAL TRIAL: NCT02490956
Title: Diagnostic Immunization With Rabies Vaccine in Patients With Primary Immunodeficiency Disorders
Brief Title: Diagnostic Immunization With Rabies Vaccine in Patients With PID
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Narissara Suratannon, Faculty of Medicine, Chulalongkorn university, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RabiesPID
Record Dates: First submitted 2015-03-30; First posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Primary Immunodeficiency
Keywords: Diagnostic immunization with rabies vaccine; Primary immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rabies vaccination (Experimental): * Verorab® (PVRV; Purified Vero Cell Vaccine) 0.5 ml intramuscular
  * Standard intramuscular regimen: ESSEN on days 0, 3, 7, 14, 28 and booster at 1 year later on days 360 and 363
  Interventions: Biological: Verorab® (PVRV; Purified Vero Cell Vaccine)

INTERVENTIONS:
Biological: Verorab® (PVRV; Purified Vero Cell Vaccine) — * Verorab® (PVRV; Purified Vero Cell Vaccine) 0.5 ml intramuscular
  * Standard intramuscular regimen: ESSEN on days 0, 3, 7, 14, 28 and booster at 1 year later on days 360 and 363

SUMMARY:
The purpose of this study is to evaluate diagnostic immunization protocol of rabies vaccine for diagnosis the patients with primary immunodeficiency disorders and study humoral and cellular immune response to rabies vaccine in patients with primary immunodeficiency.

DETAILED DESCRIPTION:
Objective Primary objective

: To study diagnostic immunization protocol of rabies vaccine for diagnosis the patients with primary immunodeficiency disorders. Secondary objective

* To study humoral and cellular immune response to rabies vaccine in patients with primary immunodeficiency.
* To study anti-rabies immunization protocol in patients with primary immunodeficiency disorders.

Population Case group: Twenty primary immunodeficiency disease patients that are diagnosed, treated and followed at Allergy and Immunology unit, Department of Pediatrics, Faculty of Medicine, Chulalongkorn University.

Control group: Twenty healthy subjects who have no underlying disease and age-matched with case patients. Inclusion and exclusion criteria

Vaccine :

* Verorab® (PVRV; Purified Vero Cell Vaccine) 0.5 ml intramuscular
* Standard intramuscular regimen: ESSEN on days 0, 3, 7, 14, 28 and booster at 1 year later on days 360 and 363

Immunological evaluations :

1. Humoral immune response :

   on 5 ml blood samples will be collected for antibody determination days 0, 14, 28, 90, 360, 367 and 374. Neutralizing antibodies will be determined blindly using the rapid fluorescent focus inhibition test (RFFIT) at Queen Saovabha Memorial Institute. Rabies neutralizing antibody will be reported in IU/ml The protective antibody level are defined rabies neutralizing antibody ≥ 0.5 IU/ml .
2. Cellular mediated immune response :

On 5 ml blood samples will be collected for antibody determination days 14, 28, 90, 360, 367 and 374. Lymphocyte proliferation response to rabies antigen will be determined by using 3H-thymidine incorporation assay.

The responder criteria are defined as stimulation index (SI index) ≥ 2.0 was considered as evidence of antigen-induced lymphocyte proliferation.

ELIGIBILITY:
Inclusion Criteria:

* Case group

  1. Patient with primary immunodeficiency diseases who follows up at Division of pediatric allergy and immunology unit, King Chulalongkorn Memorial Hospital
  2. Subject or father/mother/legally acceptable representative properly informed about the study and having signed the informed consent form.
  3. Subject is able to comply with the follow-up schedule of the protocol
* Control group

  1. Subject is healthy (from history and physical examination)
  2. Subject do not has underlying diseases.
  3. Subject do not has primary and secondary immunodeficiency diseases
  4. Subject is not receiving immunosuppressive therapy or cytotoxic drugs
  5. Subject or father/mother/legally acceptable representative properly informed about the study and having signed the informed consent form.
  6. Subject is able to comply with the follow-up schedule of the protocol
  7. Age more than 12 month old to 60 years old

Exclusion Criteria:

1. Reported history of previous rabies immunization or Rabies neutralizing antibody (Rabies Nab) > 0.5 IU/ml
2. Subject is unable to comply with the follow-up schedule of the protocol
3. Pregnancy
4. Body temperature more than 38 degree celcius at screening visit

Ages: 12 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Rabies neutralizing antibody titer (RFFIT test) | 1 year

SECONDARY OUTCOMES:
Lymphocyte proliferation response to rabies antigen (3H-Thymidine incorporation assay) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Narissara - Suratannon, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Division of Allergic and Immunology , Department of Pediatrics, Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand